CLINICAL TRIAL: NCT04507022
Title: A Randomized Controlled Study to Compare the Outcome of Two Protocols Used to Prepare the Endometrium for Frozen Embryo Transfer
Brief Title: The Outcome of Two Protocols Used to Prepare Endometrium for Frozen Embryo Transfer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rahem Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFC041120190008
Record Dates: First submitted 2020-08-01; First posted 2020-08-10 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2020-10

CONDITIONS: Infertility; Infertility, Female; Infertility, Male
MeSH Terms: conditions — Infertility; Infertility, Female; Infertility, Male | interventions — Estradiol; Progesterone; Aromatase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRT Plus Aromatase Inhibitor (Experimental): Hormone replacement treatment (HRT) will be used in all cases. Exogenous estradiol will be started on day 2 or 3 of the cycle. In all participants, 2 mg oral estradiol valerate, will be administered three times daily. Ultrasound evaluation of endometrium will be performed 10 to 12 days after starting E2. Trilaminar endometrium of 9 mm will be the targeted cutoff . If not yet ready, E2 supplementation will be continued with serial US assessment until the desired cutoff is achieved. Thereafter, participants will be randomized to two groups:
  Group A (HRT plus AI): will be given aromatase inhibitor for 5 days only (2.5 mg twice daily), along with the oral 6 mg E2. Then, daily intramuscular (IM) P in oil (100 mg IM P) will be started in addition to the daily dose of oral 6 mg E2.
  In both groups, embryos will be warmed on the 6th day of P supplementation. Before undergoing FET, endometrial thickness will be re-evaluated. IM P and 6mg E2 will be continued thereafter.
  Interventions: Drug: Estradiol Valerate; Drug: Progesterone; Drug: Aromatase inhibitor
- HRT Only (Active Comparator): Hormone replacement treatment (HRT) will be used in all cases. Exogenous estradiol will be started on day 2 or 3 of the cycle. In all participants, 2 mg oral estradiol valerate, will be administered three times daily. Ultrasound evaluation of endometrium will be performed 10 to 12 days after starting E2. Trilaminar endometrium of 9 mm will be the targeted cutoff . If not yet ready, E2 supplementation will be continued with serial US assessment until the desired cutoff is achieved. Thereafter, participants will be randomized to two groups Group B (HRT only): will be administered daily intramuscular (IM) P in oil (100 mg IM P) in addition to the daily dose of oral 6 mg E2.
  In both groups, embryos will be warmed on the 6th day of P supplementation. Before undergoing FET, endometrial thickness will be re-evaluated. IM P and 6mg E2 will be continued thereafter.
  Interventions: Drug: Estradiol Valerate; Drug: Progesterone

INTERVENTIONS:
Drug: Estradiol Valerate — 2mg three times daily
Drug: Progesterone — 100 mg daily intramuscular
Drug: Aromatase inhibitor — 2.5 mg twice daily for 5 days
  Arms: HRT Plus Aromatase Inhibitor

SUMMARY:
This is a RCT to test the outcome of two protocols used for preparation of the endometrium for frozen blastocyst embryo transfer

DETAILED DESCRIPTION:
Receptive endometrium and a good quality embryo at the blastocyst developmental stage are prerequisites for a successful implantation to occur. Blastocyst freezing techniques and survival have witnessed huge improvements in the last years. Trials to improve the outcome of frozen embryo transfer (FET) are not to be stopped. The transfer of a good quality blastocyst represents a vital part of the process. Optimization of endometrial receptivity and implantation is an everlasting challenge.

Hormone replacement therapy (HRT) is now proven to be successful for preparation of the endometrium to receive the vitrified warmed embryos. Most HRT protocols give estradiol (E2) first to reach a satisfactory endometrial thickness, then followed by progesterone to mimic the natural cycles. E2 is mostly given for 10 to 14 days and this duration might be prolonged to reach a satisfactory endometrial thickness without adversely affecting the outcome. Trans-vaginal ultrasound assessment of the endometrial thickness before the start of P supplementation has been traditionally used to predict FET cycle outcome. Clinical pregnancy rates (CPR) and live birth rates (LBR) were found to decrease for each millimetre of endometrial thickness below 7 mm. Endometrial thickness however of 9 mm was reported to be among major factors affecting LBR after FET in a large set of data.

Further, there is a recent concept that endometrial compaction (decreased thickness) between the end of estrogen phase and the day of ET has favorable impact on the outcome of FET. Different modalities were proposed to enhance endometrial compaction. One of these modalities was to decrease the dose of estrogen so as to change the estrogen- progesterone ratio as well as help in preventing further endometrial growth.

Aromatase inhibitor (AI) can be used to decrease estrogen before starting P supplementation. Additionally, there were also reports that their use had been associated with improved implantation. It appears interesting to combine the easy scheduled HRT protocol with aromatase inhibitor to maximize FET outcome.

This proposed protocol has not been tested before. In current study, HRT plus AI will be compared with HRT only. In both groups, daily intramuscular P will be given for luteal support as it was shown to give the highest ongoing pregnancy rate in FET cycles.

We did a secondary follow up analysis of some exploratory outcomes (not preregistered). These outcomes were analyzed after publication and they include Live birth rate, implantation rate, hypertensive disorders of pregnancy, large for gestation and congenital anomalies. The results of these outcomes are planned to be presented elsewhere. For openness and transparency, we felt the importance to report this follow up in the registry.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria:

* Women aged from18 - 37 years old undergoing FET using good quality blastocysts vitrified on day 5(3 BB and more) (according to Gardner and Schoolcraft 1999) (8).
* Participants having at least one good quality blastocyst (3BB and more) available for transfer after warming.
* Participants having trilaminar endometrium of 9 mm after E2 preparation.

Exclusion Criteria:

* Women younger than 18 or older than 37 years old.
* Women who have uterine abnormality or pathology.
* Women who will not meet the inclusion criteria.
* Women who will refuse to participate in in the study.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Ongoing Pregnancy Rate | at 12 weeks of gestation
  visualization of fetal cardiac pulsation by ultrasound

SECONDARY OUTCOMES:
endometrial compaction | from the end of estradiol phase to the day of embryo transfer up to 11 days
  change in endometrial thickness
clinical pregnancy rate | 6 weeks gestation
  visualization of fetal cardiac pulsation by ultrasound
Live birth rate | 24 weeks
  The birth of at least one newborn that exhibits any sign of life
Implantation rate | 6 weeks gestation
  The number of gestational sacs observed divided by the number of embryos transferred expressed as a percentage, %
Number of participants with Hypertensive disorders of pregnancy | 20 weeks gestation till postpartum
  gestational hypertension or preeclampsia
Number of participants with Large for gestational age | from gestation till delivery]
  A birth weight greater than the 90th centile of the sex-specific birth weight for a given gestational age reference.
Rate of Congenital anomalies | during pregnancy and after birth (one month after birth)
  Structural or functional disorders that occur during intra-uterine life and can be identified prenatally, at birth or later in life.

CONTACTS AND LOCATIONS:
Locations (1):
- Rahem Fertility Center, Zagazig, Sharqia Province, Egypt

REFERENCES:
- [Background] Mackens S, Santos-Ribeiro S, van de Vijver A, Racca A, Van Landuyt L, Tournaye H, Blockeel C. Frozen embryo transfer: a review on the optimal endometrial preparation and timing. Hum Reprod. 2017 Nov 1;32(11):2234-2242. doi: 10.1093/humrep/dex285. PMID 29025055
- [Background] Sekhon L, Feuerstein J, Pan S, Overbey J, Lee JA, Briton-Jones C, Flisser E, Stein DE, Mukherjee T, Grunfeld L, Sandler B, Copperman AB. Endometrial preparation before the transfer of single, vitrified-warmed, euploid blastocysts: does the duration of estradiol treatment influence clinical outcome? Fertil Steril. 2019 Jun;111(6):1177-1185.e3. doi: 10.1016/j.fertnstert.2019.02.024. Epub 2019 Apr 24. PMID 31029432
- [Background] Liu KE, Hartman M, Hartman A, Luo ZC, Mahutte N. The impact of a thin endometrial lining on fresh and frozen-thaw IVF outcomes: an analysis of over 40 000 embryo transfers. Hum Reprod. 2018 Oct 1;33(10):1883-1888. doi: 10.1093/humrep/dey281. PMID 30239738
- [Background] Pan Y, Hao G, Wang Q, Liu H, Wang Z, Jiang Q, Shi Y, Chen ZJ. Major Factors Affecting the Live Birth Rate After Frozen Embryo Transfer Among Young Women. Front Med (Lausanne). 2020 Mar 24;7:94. doi: 10.3389/fmed.2020.00094. eCollection 2020. PMID 32266278
- [Background] Haas J, Smith R, Zilberberg E, Nayot D, Meriano J, Barzilay E, Casper RF. Endometrial compaction (decreased thickness) in response to progesterone results in optimal pregnancy outcome in frozen-thawed embryo transfers. Fertil Steril. 2019 Sep;112(3):503-509.e1. doi: 10.1016/j.fertnstert.2019.05.001. Epub 2019 Jun 24. PMID 31248618
- [Background] Devine K, Richter KS, Widra EA, McKeeby JL. Vitrified blastocyst transfer cycles with the use of only vaginal progesterone replacement with Endometrin have inferior ongoing pregnancy rates: results from the planned interim analysis of a three-arm randomized controlled noninferiority trial. Fertil Steril. 2018 Feb;109(2):266-275. doi: 10.1016/j.fertnstert.2017.11.004. Epub 2018 Jan 17. PMID 29338855
- [Background] Miller PB, Parnell BA, Bushnell G, Tallman N, Forstein DA, Higdon HL 3rd, Kitawaki J, Lessey BA. Endometrial receptivity defects during IVF cycles with and without letrozole. Hum Reprod. 2012 Mar;27(3):881-8. doi: 10.1093/humrep/der452. Epub 2012 Jan 13. PMID 22246449
- [Background] Gardner DK, Schoolcraft WB. Culture and transfer of human blastocysts. Curr Opin Obstet Gynecol. 1999 Jun;11(3):307-11. doi: 10.1097/00001703-199906000-00013. PMID 10369209